CLINICAL TRIAL: NCT07163728
Title: Bone Marrow Supernatant Leptin as A Predictor of Chemotherapy Sensitivity in AML Patients
Brief Title: Leptin: A Marker for AML Chemo-Sensitivity
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AML-Leptin
Record Dates: First submitted 2025-09-02; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: AML; Adult
Keywords: AML; Leptin; Chemotherapy sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Bone marrow supernatant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Myeloid Leukemia (AML) is a malignant clonal disorder of hematopoietic stem/progenitor cells, with a five-year survival rate of approximately 30%. Chemotherapy resistance and relapse remain major challenges. Increased bone marrow adipocytes contribute to AML cell drug resistance.This study found that elevated levels of the adipokine leptin enhance oxidative phosphorylation (OXPHOS) in AML cells, accompanied by increased mitochondrial reactive oxygen species (mtROS), which stimulates antioxidant capacity and thereby induces chemotherapy resistance. By establishing a correlation between leptin levels in bone marrow supernatant and clinical outcomes in AML patients, this research provides novel strategic insights for targeting drug resistance and improving prognostic evaluation.

DETAILED DESCRIPTION:
In this prospective study, we will collect bone marrow supernatant samples from patients diagnosed with Acute Myeloid Leukemia (AML) to evaluate the levels of leptin. Our aim is to explore whether elevated leptin levels can serve as a predictive biomarker for poor treatment outcomes following standard chemotherapy regimens. The findings may help in stratifying patient risk and personalizing therapeutic approaches in AML treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis aligns with the "Chinese guidelines for diagnosis and treatment of adult acute myeloid leukemia (not APL) (2023)";
2. All patients are experiencing their first onset of the disease and have not received any related chemotherapy prior to the study;
3. Patients participate in the study accompanied by family members and sign informed consent documents.

Exclusion Criteria:

1. Patients with concurrent malignancies requiring treatment;
2. Presence of infectious diseases, including SARS, viral hepatitis, or HIV/ AIDS;
3. Major surgery performed within the last 21 days;
4. Performance Status (PS) score >3;
5. Severe liver or kidney dysfunction or serious infection;
6. Severe psychiatric conditions that impair understanding of the study protocol or voluntary withdrawal.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective study enrolls patients who fulfill the diagnostic criteria for AML (excluding APL), with an age requirement of over 18 years and no restrictions on gender. Participation is entirely voluntary, with each participant or their legal guardian being thoroughly informed about the study details and signing an informed consent form. Participants are willing to adhere to and capable of completing all required study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 month
  The primary endpoint of this study is the overall response rate (ORR) after Chemotherapy

SECONDARY OUTCOMES:
CR | 1 month
  The secondary endpoints is the complete remission (CR) rate after Chemotherapy
CRi | 1 month
  The secondary endpoints is the complete remission with incomplete blood count recovery (CRi) rate after Chemotherapy
PR | 1 month
  The secondary endpoints is the partial remission (PR) rate after Chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Huang, Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No